CLINICAL TRIAL: NCT01841944
Title: Giving Omega-3 Fatty Acids to Elderly Patients Diagnosed With Acute Myocardial Infarction to Investigate the Effect on Cardiovascular Morbidity and Mortality
Brief Title: Omega-3 Fatty Acids in Elderly Patients With Acute Myocardial Infarction
Acronym: OMEMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University Hospital, Akershus (Other); Asker & Baerum Hospital (Other); Helse Stavanger HF (Other Government)
Responsible Party: Principal Investigator, Are Annesønn Kalstad, Medical Doctor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2012/14890; 2012-004478-25 (EudraCT Number)
Record Dates: First submitted 2013-04-16; First posted 2013-04-29 (Estimated); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Myocardial Infarction; Heart Failure; Myocardial Revascularization; Atrial Fibrillation
Keywords: Fatty Acids, Omega-3; Aged; Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction; Heart Failure; Atrial Fibrillation | interventions — Pikasol; Docosahexaenoic Acids; Fatty Acids, Unsaturated; Corn Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pikasol (Active Comparator): Pikasol®, 3 capsules (1.8 g EPA+DHA)/day
  Interventions: Drug: Pikasol
- Corn oil (Placebo Comparator): 3x capsules of corn oil pr day
  Interventions: Other: Corn oil

INTERVENTIONS:
Drug: Pikasol — Pikasol®, 3 capsules (1.8 g EPA+DHA)/day
  Other Names: omega-3; polyunsaturated fatty acids
  Arms: Pikasol
Other: Corn oil — Corn oil (56% linoleic acid, 32% oleic acid, 10% palmitic acid), unchanged and according to the manufacturer
  Arms: Corn oil

SUMMARY:
The aim of the present study is to investigate the possible effects of supplementation with 1.8 g/day of n-3 polyunsaturated fatty acids on cardiovascular morbidity and mortality during a follow-up period of 2 years in an elderly population after having experienced an acute myocardial infarction.

The hypothesis is that this supplementation on top of modern therapy will reduce the combined cardiovascular end-point of death, non-fatal myocardial infarction, stroke, revascularizations or hospitalization for new or worsened heart failure with at least 30%.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute myocardial infarction discharged from hospital alive

Exclusion Criteria:

* Being part of another randomized trial
* Documented intolerance for omega-3 fatty acids
* Additional disease state that is thought to be incompatible with compliance to the study drugs
* Additional disease state thought to reduce survival for the follow-up time of 2 years

Ages: 70 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1027 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
Combined total mortality, first event of non-fatal myocardial infarction, stroke, revascularization or hospital admission for new or worsened heart failure. | 24months

SECONDARY OUTCOMES:
Occurence of new onset atrial fibrillation | 24months

CONTACTS AND LOCATIONS:
Overall Officials: Harald Arnesen, MD Phd, Study Chair — Center for Clinical Heart Research; Svein Solheim, MD phd, Study Director — Center for Clinical Heart Research; Ingebjørg Seljeflot, Phd, Study Director — Center for Clinical Heart Research; Kristian Laake, MD, Principal Investigator — Center for Clinical Heart Research; Peder Myhre, MD, Principal Investigator — Center for Clinical Heart Research; Are A Kalstad, MD, Principal Investigator — Center for Clinical Heart Research
Locations (4):
- Norway (4):
  - Asker and Bærum Hospital, Rud, Bærum
  - Akershus university hospital HF, Lørenskog
  - Oslo University Hospital(Ullevaal), Oslo
  - Stavanger University Hospital, Stavanger

REFERENCES:
- [Derived] Chiva-Blanch G, Bratseth V, Laake K, Arnesen H, Solheim S, Schmidt EB, Badimon L, Seljeflot I. One year of omega 3 polyunsaturated fatty acid supplementation does not reduce circulating prothrombotic microvesicles in elderly subjects after suffering a myocardial infarction. Clin Nutr. 2021 Dec;40(12):5674-5677. doi: 10.1016/j.clnu.2021.10.007. Epub 2021 Oct 20. PMID 34742136
- [Derived] Kalstad AA, Myhre PL, Laake K, Opstad TB, Tveit A, Solheim S, Arnesen H, Seljeflot I. Biomarkers of ageing and cardiac remodeling are associated with atrial fibrillation. Scand Cardiovasc J. 2021 Aug;55(4):213-219. doi: 10.1080/14017431.2021.1889653. Epub 2021 Mar 2. PMID 33650449
- [Derived] Kalstad AA, Myhre PL, Laake K, Tveit SH, Schmidt EB, Smith P, Nilsen DWT, Tveit A, Fagerland MW, Solheim S, Seljeflot I, Arnesen H; OMEMI Investigators. Effects of n-3 Fatty Acid Supplements in Elderly Patients After Myocardial Infarction: A Randomized, Controlled Trial. Circulation. 2021 Feb 9;143(6):528-539. doi: 10.1161/CIRCULATIONAHA.120.052209. Epub 2020 Nov 15. PMID 33191772
- [Derived] Kalstad AA, Tveit S, Myhre PL, Laake K, Opstad TB, Tveit A, Schmidt EB, Solheim S, Arnesen H, Seljeflot I. Leukocyte telomere length and serum polyunsaturated fatty acids, dietary habits, cardiovascular risk factors and features of myocardial infarction in elderly patients. BMC Geriatr. 2019 Dec 27;19(1):376. doi: 10.1186/s12877-019-1383-9. PMID 31881852
- [Derived] Laake K, Myhre P, Nordby LM, Seljeflot I, Abdelnoor M, Smith P, Tveit A, Arnesen H, Solheim S. Effects of omega3 supplementation in elderly patients with acute myocardial infarction: design of a prospective randomized placebo controlled study. BMC Geriatr. 2014 Jun 13;14:74. doi: 10.1186/1471-2318-14-74. PMID 24928284